CLINICAL TRIAL: NCT05258422
Title: Stereotactic Arrhythmia Radioablation for Ventricular Tachycardia (StAR-VT): a Single Centre, Phase II, Dose De-escalation, Non-inferiority, Clinical Trial.
Brief Title: Stereotactic Arrhythmia Radioablation for Ventricular Tachycardia (StAR-VT)
Acronym: StAR-VT
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Joanne Alfieri, Associate Professor Radiation Oncology, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-7202
Record Dates: First submitted 2022-02-09; First posted 2022-02-28 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Ventricular Tachycardia; Arrhythmia; Arrhythmic Storm; Radiation Toxicity
Keywords: stereotactic body radiotherapy, ventricular tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular; Arrhythmias, Cardiac; Radiation Injuries | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: This study will assess the non-inferiority of treatment with single fraction of 20 Gy delivered with stereotactic body radiotherapy in comparison with historical controls treated with a single fraction of 25 Gy. Based on historical controls, the investigators anticipate an incidence rate of approximately five VT events per person-year in participants treated with 25 Gy historical comparator. Based on a Poisson distribution and using a non-inferiority margin of 8.5 events per-year (corresponding to an incident rate ratio of 1.7), recruitment of nine participants will provide 80% power when using a one-sided type I error set at 0.05.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiation: 20 Gy in 1 fraction (Experimental): External beam, stereotactic body radiotherapy of 20 Gy delivered in 1 fraction to the planning target volume (PTV) of the arrhythmogenic substrate
  Interventions: Radiation: stereotactic body radiotherapy, 20 Gy in 1 fraction

INTERVENTIONS:
Radiation: stereotactic body radiotherapy, 20 Gy in 1 fraction — A single dose of focused radiation therapy of 20 Gy in 1 fraction to the PTV of the arrhythmogenic substrate
  Other Names: stereotactic ablative radiotherapy, 20 Gy in 1 fraction

SUMMARY:
In 2017 a novel treatment approach to a series of 5 patients with refractory VT was introduced, using ablative radiation with a stereotactic body radiation therapy (SBRT) technique to arrhythmogenic scar regions defined by noninvasive cardiac mapping. More recently, Robinson et al. reported on the results of their Electrophysiology-Guided Noninvasive Cardiac Radioablation for Ventricular Tachycardia (ENCORE-VT) trial, also using a similar SBRT technique in a series of 17 patients with refractory VT. Both studies report a marked reduction in VT burden, a decrease in antiarrhythmic drug use, and an improvement in quality of life. Since then, numerous other centres have detailed their initial experience with this technique. These initial results suggest that this new treatment paradigm has the potential to improve morbidity and mortality for patients suffering from treatment-refractory VT by means of a minimally invasive technique, but requires further validation for widespread use.

The appropriate dose for therapeutic effect of this new treatment is not well established as only a single dose prescription of 25 Gy in 1 fraction has been described with benefit. In this phase 2 trial, the investigators plan on expanding the experience with this technique but also by contributing to understanding the relationship between dose-effect relationship through a dose de-escalation stratification, to 20 Gy in 1 fraction, with the goal of minimizing possible adverse events and radiation dose to surrounding healthy tissue while maintaining a clinical benefit.

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) is a potentially life-threatening arrhythmia characterized by electrical re-entry within patches of heterogeneous myocardial fibrosis leading to sustained consecutive ventricular beats at a rate > 100 per minute. VT is classified based on hemodynamic stability, duration (less than or greater than 30 seconds), morphology (monomorphic or polymorphic), and mechanism (scar-related re-entry, automaticity, triggered activity.

In patients with monomorphic VT, implantable cardioverter-defibrillators (ICDs) have become the cornerstone of therapy in decreasing mortality, through the prevention of sudden death from potentially lethal sustained arrhythmia in select patients. However, ICDs have no effect on the underlying arrhythmogenic substrate or fibrotic scar and thus are primarily a symptom-control therapy; patients may develop recurrent and debilitating shocks associated with an increase in mortality. Currently, catheter ablation (CA) for VT is used as an adjunctive therapy for patients who are refractory to medical therapy. A recent systematic review and meta-analysis of randomized controlled trials and observation studies comparing medical therapy and catheter ablation for VT shows that CA is superior to medical therapy for scar-related VT with respect to VT recurrence and the life-threatening VT storm. Despite this, there is still a high reported incidence of VT recurrence in both medically-treated (48%) and ablation-treated (39%) patients, suggesting that the current treatment paradigm is suboptimal for good control of this debilitating arrhythmia.

In 2017, Cuculich et al. introduced a novel treatment approach to a series of 5 patients with refractory VT, using ablative radiation with a stereotactic body radiation therapy (SBRT) technique to arrhythmogenic scar regions defined by noninvasive cardiac mapping. More recently, Robinson et al. reported on the results of their Electrophysiology-Guided Noninvasive Cardiac Radioablation for Ventricular Tachycardia (ENCORE-VT) trial, also using a similar SBRT technique in a series of 17 patients with refractory VT. Both studies report a marked reduction in VT burden, a decrease in antiarrhythmic drug use, and an improvement in quality of life. These initial results suggest that this new treatment paradigm has the potential to vastly improve morbidity and mortality for patients suffering from VT by means of a minimally invasive technique, but requires further validation for widespread use.

Additionally, the appropriate dose for therapeutic effect of this new treatment is not well established as only a single dose prescription of 25 Gy in 1 fraction has been described with benefit. In this phase 2 trial, the investigators plan on expanding the experience with this technique but also by contributing to understanding the relationship between dose-effect relationship through a dose de-escalation stratification, to 20 Gy in 1 fraction, with the goal of minimizing possible adverse events and radiation dose to surrounding healthy tissue while maintaining a clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Ishemic or non-ischemic cardiomyopathy
* Recurrent episodes of monomorphic ventricular tachycardia having failed standard treatment with at least 1 antiarrhythmic drug
* Previous endocardial and/or epicardial electrophysiology study and ablation.

Participants who have a contraindication to electrophysiology studies (ventricular thrombus, absence of vascular access, valvular heart disease or mechanical heart valve that precludes left-ventricular access) may be eligible for the protocol provided the arrhythmic substrate can be defined through non-invasive methods.

Exclusion Criteria:

* Previous RT in the treatment field that precludes furth RT
* Active connective tissue disease
* Interstitial pulmonary fibrosis
* Pregnant or breastfeeding individuals
* Participants who plan to become pregnant or breast feed during the study duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in arrhythmia burden measured by the number of VT events | 6 months and 12 months following study intervention
  Changes in arrhythmia burden measured by the number of VT events comparing the 12-month period after a single fraction of 20 Gy SBRT with a single fraction of 25 Gy in historical controls
Change in arrhythmia burden measured by the number of ICD events | 6 months and 12 months following study intervention
  Changes in arrhythmia burden measured by the number of ICD events comparing the 12-month period after a single fraction of 20 Gy SBRT with a single fraction of 25 Gy in historical controls
Acute radiation toxicity within the first 90 days measured by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 90 days following study intervention.
  Rate of severe adverse events at less than or equal to 90 days that were treatment related (possibly, probably, or definitely) as defined using the CTCAE v5.0

SECONDARY OUTCOMES:
Late radiation toxicity occurring after the first 90 days until 5 years measured by the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 90 days - 5 years following study intervention
  Severe adverse events as defined by CTCAE v5.0 occuring after the first 90 days following treatment
Changes in number and doses of antiarrhythmic drugs | 1 year, 3 years, and 5 years following study intervention
  Changes in number and doses of all antiarrhythmic drugs that are used before and in the 5 year follow-up after the study intervention
Patient-Reported Quality of life as measured by the short form-36 questionnaire | 6 months, 1 year, 3 years, and 5 years following study intervention
  Patient-Reported Quality of life as measured by the short form-36 questionnaire
Patient-Reported Quality of life as measured by the Arrhythmia-specific questionnaire in Tachycardia and arrhythmia (ASTA) | 6 months, 1 year, 3 years, and 5 years following study intervention
  Patient-Reported Quality of life as measured by the Arrhythmia-specific questionnaire in Tachycardia and arrhythmia (ASTA)

OTHER OUTCOMES:
Overall Survival | 5 years following radiation therapy
  The overall survival of participants following the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Alfieri, MD, Principal Investigator — MUHC division of radiation oncology/RIMUHC; Martin L Bernier, MD, Principal Investigator — MUHC division of cardiology
Locations (1):
- Cedars Cancer Center, McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
available upon request

REFERENCES:
- [Background] AlKalbani A, AlRawahi N. Management of monomorphic ventricular tachycardia electrical storm in structural heart disease. J Saudi Heart Assoc. 2019 Jul;31(3):135-144. doi: 10.1016/j.jsha.2019.05.001. Epub 2019 May 11. PMID 31198398
- [Background] Shenthar J. Unusual Incessant Ventricular Tachycardia: What Is the Underlying Cause and the Possible Mechanism? Circ Arrhythm Electrophysiol. 2015 Dec;8(6):1507-11. doi: 10.1161/CIRCEP.115.002886. No abstract available. PMID 26671936
- [Background] Anderson RD, Ariyarathna N, Lee G, Virk S, Trivic I, Campbell T, Chow CK, Kalman J, Kumar S. Catheter ablation versus medical therapy for treatment of ventricular tachycardia associated with structural heart disease: Systematic review and meta-analysis of randomized controlled trials and comparison with observational studies. Heart Rhythm. 2019 Oct;16(10):1484-1491. doi: 10.1016/j.hrthm.2019.05.026. Epub 2019 May 29. PMID 31150816
- [Background] Hohnloser SH, Kuck KH, Dorian P, Roberts RS, Hampton JR, Hatala R, Fain E, Gent M, Connolly SJ; DINAMIT Investigators. Prophylactic use of an implantable cardioverter-defibrillator after acute myocardial infarction. N Engl J Med. 2004 Dec 9;351(24):2481-8. doi: 10.1056/NEJMoa041489. PMID 15590950
- [Background] Aziz Z, Tung R. Novel Mapping Strategies for Ventricular Tachycardia Ablation. Curr Treat Options Cardiovasc Med. 2018 Mar 23;20(4):34. doi: 10.1007/s11936-018-0615-1. PMID 29572643
- [Background] Cuculich PS, Schill MR, Kashani R, Mutic S, Lang A, Cooper D, Faddis M, Gleva M, Noheria A, Smith TW, Hallahan D, Rudy Y, Robinson CG. Noninvasive Cardiac Radiation for Ablation of Ventricular Tachycardia. N Engl J Med. 2017 Dec 14;377(24):2325-2336. doi: 10.1056/NEJMoa1613773. PMID 29236642
- [Background] Robinson CG, Samson PP, Moore KMS, Hugo GD, Knutson N, Mutic S, Goddu SM, Lang A, Cooper DH, Faddis M, Noheria A, Smith TW, Woodard PK, Gropler RJ, Hallahan DE, Rudy Y, Cuculich PS. Phase I/II Trial of Electrophysiology-Guided Noninvasive Cardiac Radioablation for Ventricular Tachycardia. Circulation. 2019 Jan 15;139(3):313-321. doi: 10.1161/CIRCULATIONAHA.118.038261. PMID 30586734
- [Background] Walfridsson U, Arestedt K, Stromberg A. Development and validation of a new Arrhythmia-Specific questionnaire in Tachycardia and Arrhythmia (ASTA) with focus on symptom burden. Health Qual Life Outcomes. 2012 Apr 30;10:44. doi: 10.1186/1477-7525-10-44. PMID 22545926
- [Background] Knutson NC, Samson PP, Hugo GD, Goddu SM, Reynoso FJ, Kavanaugh JA, Mutic S, Moore K, Hilliard J, Cuculich PS, Robinson CG. Radiation Therapy Workflow and Dosimetric Analysis from a Phase 1/2 Trial of Noninvasive Cardiac Radioablation for Ventricular Tachycardia. Int J Radiat Oncol Biol Phys. 2019 Aug 1;104(5):1114-1123. doi: 10.1016/j.ijrobp.2019.04.005. Epub 2019 Apr 16. PMID 31002942
- [Background] Duane F, Aznar MC, Bartlett F, Cutter DJ, Darby SC, Jagsi R, Lorenzen EL, McArdle O, McGale P, Myerson S, Rahimi K, Vivekanandan S, Warren S, Taylor CW. A cardiac contouring atlas for radiotherapy. Radiother Oncol. 2017 Mar;122(3):416-422. doi: 10.1016/j.radonc.2017.01.008. Epub 2017 Feb 21. PMID 28233564
- [Background] Hanna GG, Murray L, Patel R, Jain S, Aitken KL, Franks KN, van As N, Tree A, Hatfield P, Harrow S, McDonald F, Ahmed M, Saran FH, Webster GJ, Khoo V, Landau D, Eaton DJ, Hawkins MA. UK Consensus on Normal Tissue Dose Constraints for Stereotactic Radiotherapy. Clin Oncol (R Coll Radiol). 2018 Jan;30(1):5-14. doi: 10.1016/j.clon.2017.09.007. Epub 2017 Oct 13. PMID 29033164
- [Background] Desai MY, Windecker S, Lancellotti P, Bax JJ, Griffin BP, Cahlon O, Johnston DR. Prevention, Diagnosis, and Management of Radiation-Associated Cardiac Disease: JACC Scientific Expert Panel. J Am Coll Cardiol. 2019 Aug 20;74(7):905-927. doi: 10.1016/j.jacc.2019.07.006. PMID 31416535
- [Background] Pinta C, Besse R. Stereotactic ablative body radiotherapy for ventricular tachycardia: An alternative therapy for refractory patients. Anatol J Cardiol. 2021 Dec;25(12):858-862. doi: 10.5152/AnatolJCardiol.2021.187. PMID 34866579
- [Background] Gerard IJ, Bernier M, Hijal T, Kopek N, Pater P, Stosky J, Stroian G, Toscani B, Alfieri J. Stereotactic Arrhythmia Radioablation for Ventricular Tachycardia: Single Center First Experiences. Adv Radiat Oncol. 2021 Apr 20;6(4):100702. doi: 10.1016/j.adro.2021.100702. eCollection 2021 Jul-Aug. No abstract available. PMID 34095614
- [Background] Lee J, Bates M, Shepherd E, Riley S, Henshaw M, Metherall P, Daniel J, Blower A, Scoones D, Wilkinson M, Richmond N, Robinson C, Cuculich P, Hugo G, Seller N, McStay R, Child N, Thornley A, Kelland N, Atherton P, Peedell C, Hatton M. Cardiac stereotactic ablative radiotherapy for control of refractory ventricular tachycardia: initial UK multicentre experience. Open Heart. 2021 Nov;8(2):e001770. doi: 10.1136/openhrt-2021-001770. PMID 34815300
- [Background] Chiu MH, Mitchell LB, Ploquin N, Faruqi S, Kuriachan VP. Review of Stereotactic Arrhythmia Radioablation Therapy for Cardiac Tachydysrhythmias. CJC Open. 2020 Nov 13;3(3):236-247. doi: 10.1016/j.cjco.2020.11.006. eCollection 2021 Mar. PMID 33778440
- [Background] Sharma A, Wong D, Weidlich G, Fogarty T, Jack A, Sumanaweera T, Maguire P. Noninvasive stereotactic radiosurgery (CyberHeart) for creation of ablation lesions in the atrium. Heart Rhythm. 2010 Jun;7(6):802-10. doi: 10.1016/j.hrthm.2010.02.010. Epub 2010 Feb 13. PMID 20156591
- [Background] Blanck O, Bode F, Gebhard M, Hunold P, Brandt S, Bruder R, Grossherr M, Vonthein R, Rades D, Dunst J. Dose-escalation study for cardiac radiosurgery in a porcine model. Int J Radiat Oncol Biol Phys. 2014 Jul 1;89(3):590-8. doi: 10.1016/j.ijrobp.2014.02.036. Epub 2014 Apr 18. PMID 24751407
- [Background] Amino M, Yoshioka K, Fujibayashi D, Hashida T, Furusawa Y, Zareba W, Ikari Y, Tanaka E, Mori H, Inokuchi S, Kodama I, Tanabe T. Year-long upregulation of connexin43 in rabbit hearts by heavy ion irradiation. Am J Physiol Heart Circ Physiol. 2010 Mar;298(3):H1014-21. doi: 10.1152/ajpheart.00160.2009. Epub 2010 Jan 8. PMID 20061548
- See also: CTCAE v5.0 — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm